CLINICAL TRIAL: NCT02578264
Title: Molecular Stethoscope for Colon Cancer Detection
Brief Title: Molecular Stethoscope
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Sequenom, Inc. (Industry)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute, Scripps Translational Science Institute
Other Study IDs: 15-6616
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: All subjects enrolled in the study will provide tumor and normal tissue and blood samples.

SUMMARY:
The study aims to provide a more complete characterization and understanding of the genetic causes of and tumor DNA detection potential in colorectal cancer. Ultimately findings of this study will be used to develop early detection tests for colorectal cancer that are minimally invasive (based on a blood test). It is hoped that reliable, minimally invasive, early detection methods will lead to improved screening rates, increased screening safety, longer colorectal cancer survival, and overall cost savings.

In order to assess the test's ability to detect tumor DNA, 25 participants with known colorectal cancer who will be undergoing surgical resection of the colon as part of their clinical care will be recruited. The investigators will collect blood from participants prior to surgery, tumor and normal tissue removed during surgery, a series of blood samples after surgery for up to one year and relevant medical records. DNA variants identified in blood will be compared against tissue samples. Serial samples will be analyzed to assess the variance in amount of circulating tumor DNA across time with standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer sent for surgical colonic resection (all stages) OR
* High risk adenoma sent for surgical colonic resection

Exclusion Criteria:

* Chemotherapy before surgical treatment
* Invasive procedure resulting in damage to tissue (e.g., surgery, biopsy, thermal ablation) in the 7 days prior to baseline (pre-surgical) blood collection
* Radiation therapy before surgical treatment
* Bone marrow transplant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer that will be receiving surgical removal of their cancer as part of their care.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Determining sensitivity of assay in known cancer patients | 2 years
  The sensitivity (% positive out of all diseased patients) of circulating tumor DNA detection from the blood samples will be calculated against the gold standard of surgical pathology reports in this pilot group of patients with known colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Topol, MD, Principal Investigator — Scripps Translational Science Institute